CLINICAL TRIAL: NCT01919021
Title: Pilot Study: Assessment of Gastric Motor and Sensory Function to a Mixed Liquid and Solid Test Meal by Gamma Scintigraphy, Magnetic Resonance Imaging and a Nutrient Drink Test in Health and Patients With Disorders of Gastric Function
Brief Title: Assessment of Gastro-Intestinal Function to a Mixed Meal by Non-invasive Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11GA006
Record Dates: First submitted 2013-07-10; First posted 2013-08-08 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Functional Dyspepsia; Diabetic Gastroparesis
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Sensation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Magnetic Resonance Imaging MRI — 400ml of milkshake and 12 agar beads are ingested and gamma scintigraphy scanning completed to document gastric emptying and outcome measures listed earlier.
Other: Gamma Scintigraphy — 400ml of milkshake and 12 agar beads are ingested and gamma scintigraphy scanning completed to document gastric emptying and outcome measures listed earlier.
Procedure: Assessment of Gastric motor and sensory function

SUMMARY:
Dyspeptic symptoms, such as pain after eating, bloating and nausea all have major impact on quality of life and health care costs. When no structural cause is identified, patients are diagnosed with functional dyspepsia. This trial aims to identify objective abnormalities of stomach function that explain patient's symptoms and establish diagnosis. Another group are diabetic patients who can often develop similar symptoms, labelled as diabetic gastroparesis. In some cases this is associated with delayed gastric emptying but not all.

24 patients with functional dyspepsia will be studied and 24 healthy controls (to establish normal ranges) and 24 diabetic patients with symptoms of functional dyspepsia.

The utility of 3 different non-invasive investigations will be assessed. At screening the nutrient drink test (NDT) asks the patient to drink 40ml of milkshake (0.75kcal/ml) every minute and score symptoms every 5 minutes. The patient continues until they reach the maximum tolerated volume.

Participants will then be randomized to undergo non-invasive imaging on two separate test days by magnetic resonance imaging (MRI) and gastric scintigraphy MRI will be completed with the patient ingesting 400ml of milkshake (identical to NDT) and 12 agar beads (no additional calories) of known breaking strength. The emptying of the stomach will be visualised with the MRI alongside symptom recording.

Gamma scintigraphy will ingest the same meal as for the MRI scan but radioactive labelling will allow the rate of liquid and solid meal emptying to be visualised alongside symptom recording.

Additionally, blood sugars will be recorded before nutrient drink test and at 15 and 30 minutes following ingestion of 400ml of milkshake and 12 agar beads.

Data will be analyzed to assess the association of objective abnormalities of gastric function and patient symptoms. Additionally the results of non-invasive imaging by MRI and GS will be compared to assess the optimal measurement of gastric function and emptying in this clinical scenario.

ELIGIBILITY:
Inclusion Criteria:

1. Be an adult patient above 18 years old
2. Have a body mass index of >18 and <30kg.m2 and not exceed a waist circumference of 99cm at 5cm above ileal crest
3. Be able to give voluntary informed consent and from whom written consent to participate has been obtained.
4. Be able to understand the study, willing to co-operate with the study procedures and able to attend all study assessments.
5. Be willing to abstain from alcohol for 24 hours before and during the imaging appointment.
6. Be willing to fast from midnight prior to the screening and imaging appointment
7. Be able to ingest at least 400ml nutrient liquid (0.75kcal/ml at 40ml/min) during a Nutrient Drinking Test without experiencing more than moderate dyspeptic symptoms (no such restriction for patients with dyspeptic symptoms)
8. Be able to swallow a solid agar bead between 7.5 and 11.5 mm in diameter
9. Be willing to consent to their General Practitioner (GP) being informed of their participation.

Exclusion Criteria:

1. Have a history of gastrointestinal disease or surgery (other than appendicitis or hysterectomy)
2. Have ongoing disease requiring active management (including impaired renal clearance GFR <50 mL/min/1.73 m2)
3. Have a documented history of alcohol or drug abuse
4. Fail to satisfy the investigator's assessment of fitness to participate based on a survey of inclusion and exclusion criteria
5. Have consumed alcohol within 24 hours of start of study
6. Have participated in a similar study involving the use of radioisotopes in the previous 3 months such that participating in the current study would exceed the recommended yearly exposure limit (5mSv)
7. Take any medication which may affect oesophageal or gastric motility for a minimum 7 days
8. Have had previous history of gastric surgery
9. Have active upper gastrointestinal diseases
10. Have an active Eating Disorder
11. Have an allergy to milk protein (milk based, lactose free test meal)
12. Be a vegan
13. Be pregnant or breastfeeding
14. Have any contraindication to MRI scanning according to local guidelines

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Maximum volume ingested at nutrient drink test (ml) | Study Day
  Maximum of milkshake ingested at maximum satiety
Gastric emptying rate (ml/min) for liquids | Study day
  gastric emptying rate measured by non-invasive imaging
Gastric emptying rate (ml/min) for solids | Study Day
  Gastric emptying rate measured by non-invasive imaging
Time taken for 50% gastric emptying (T50, minutes) for liquids | Study day-After 50% of contents of stomach has emptied
  time taken for 50% of gastric contents to leave the stomach
Time take for 50% gastric emptying (T50, minutes) solids | Study day-after 50% of contents of stomach has emptied
  Time taken for 50% of gastric contents to leave the stomach

SECONDARY OUTCOMES:
Sensation at 200ml, 400ml and at completion of nutrient drink test (fullness, bloating, nausea, heartburn, epigastric pain) | Study day
  Visual analogue score for each sensation (score up to 100 points)
Glycaemic response at 15 minutes and 30 minutes post 400ml milkshake | study day
  Blood glucose (mmol/l)
Gastric volume at 200ml nutrient ingestion | Study day
  Measurement of gastric volume (ml) on MRI and gamma scintigraphy
Gastric volume at 400ml nutrient ingestion | study day
  measurement of gastric volume (ml) on MRI and gamma scintography
Gastric contractile wave contractile frequency | study day
  contractile frequency within stomach
Oro-caecal Transit time | study day
  Time taken for 50% gastric contents to enter caecum
Sensation threshold volume for fullness, bloating, nausea, heartburn and epigastric pain | study day
  Gastric volume recorded at time of maximum symptom scores
Sensation at 200ml and 400ml ingestion of test meal (fullness, bloating, nausea, heartburn, epigastric pain) | study day
  Visual analogue score for each sensation (score up to 100 points)
GI Hormone Assessment | Study day
  5 ml of blood will be taken at time 0, 30, 60 and 120 min. GI peptide hormones will then be analysed from the samples.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fox, BMBS, MD, Principal Investigator — University of Nottingham
Locations (1):
- National Institute of Health Research Biomedical Research Unit, Nottingham Digestve Diseases Centre, University of Nottingham,, Nottingham, United Kingdom